CLINICAL TRIAL: NCT06289972
Title: Development, Validity and Reliability of a Caregiver Version of the Breathlessness Beliefs Questionnaire
Brief Title: Development,Validity and Reliability of a Caregiver Version of the Breathlessness Beliefs Questionnaire
Status: Completed | Type: Observational
Sponsor: Halic University (Other)
Responsible Party: Principal Investigator, Seda Saka, Asst. Prof., Halic University
Other Study IDs: HUvbayraktaroglu1
Record Dates: First submitted 2024-02-26; First posted 2024-03-04 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Cystic Fibrosis; Parents
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this methodological study is to determine the reliability and validity of the The Breathlessness Beliefs Questionnaire Caregiver Version (BBQ-C) version in assessing dysfunctional breathlessness beliefs in caregivers of children with cystic fibrosis.

DETAILED DESCRIPTION:
Cystic fibrosis (CF) is an inherited disease characterized by pulmonary involvement. Children with CF may have obstructive lung disease and related dyspnea, which may progress to respiratory failure and mortality. Dyspnea may lead to activity limitation. Parents who take care of children with CF may be protective of their children's social environment for some reasons such as the risk of infection. The Breathlessness Beliefs Questionnaire (BBQ) is a Turkish validated scale developed to assess dysfunctional beliefs about dyspnea. Based on the idea that parents may develop dysfunctional dyspnea belief behavior in their children with CF, the aim of this study was to develop a caregiver version of the BBQ (The Breathlessness Beliefs Questionnaire Caregiver Version-BBQ-C) and to investigate the validity and reliability of the scale in assessing dysfunctional dyspnea beliefs in parents of children with CF.

ELIGIBILITY:
Inclusion Criteria:

* To be between 25-75 years old,
* To be literate in Turkish,
* Being a mother, father or other caregiver of a child,
* Voluntarily agreeing to participate in the study,
* Be taking care of the child for at least one year

Exclusion Criteria:

* Having cognitive impairment at a level that prevents cooperation with the scales,
* Not living in the same household with a child with cystic fibrosis.

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population of the study will consist of parents of CF patients who come to the Pediatric Chest Diseases Outpatient Clinic of a private hospital for routine control. The sample will consist of parents who fulfill the inclusion and exclusion criteria and volunteer to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2024-02-20 (Actual); Primary Completion 2024-07-11 (Actual); Study Completion 2024-07-11 (Actual)

PRIMARY OUTCOMES:
The Breathlessness Beliefs Questionnaire (Caregiver Version) (BBQ-C) | baseline, after 15 days
  The BBQ-C will assess dysfunctional dyspnea beliefs in caregivers.The questionnaire has a minimum score of 11 and a maximum score of 55. As the total score increases, the belief in dysfunctional dyspnea increases.

SECONDARY OUTCOMES:
Cystic Fibrosis Questionnaire Revised (CFQ-R) for parent version | baseline, after 15 days
  The CFQ-R assesses quality of life. The CFQ-R is a cystic fibrosis-specific scale developed separately for both the child and the parent. The parent version consists of 50 items. Scores for each HRQoL domain; after recoding, each item is summed to generate a domain score and standardized. Scores range from 0 to 100, with higher scores indicating better health. CD-Rom Program available for scoring the CFQ-R.
Parent Attitude Scale (PAS) | baseline, after 15 days
  The PAS is assess to perceived parental attitude according to child.The scale has three sub-dimensions: acceptance/affection, control/supervision and psychological autonomy. Accordingly, since the scale is scored as Always 5; Mostly 4; No opinion 3; Occasionally 2; Never 1, the individual to whom the scale is applied receives a minimum score of 15 and a maximum score of 75 from each dimension separately. Each dimension is evaluated according to whether the scores are low or high. In whichever dimension the score is higher, it is accepted that the child perceives parental attitude in that way.
Perceived Social Support Scale (PSS) | baseline, after 15 days
  The PSS is assess to perceived social support according to child. The scale includes 5 items on social support perceived from mother and 5 items on social support perceived from father, and 4 items on social support perceived from peers. A minimum of 14 points and a maximum of 70 points can be obtained from the scale. As the total score increases, the child's perception of social support increases.
Parent Attitude Scale | baseline, after 15 days
  Parent Attitude Scale is assess to perceived parental attitude according to parent. Democratic (17 items), Authoritarian (11 items), Overprotective (9 items), Permissive (9 items). In scoring, scores and corresponding responses were 5 for "always", 4 for "most of the time", 3 for "sometimes", 2 for "rarely" and 1 for "never". Having a high score meant to adopt the behavior style represented by that domain.

CONTACTS AND LOCATIONS:
Locations (1):
- Haliç University, Istanbul, Eyup, Turkey (Türkiye)